CLINICAL TRIAL: NCT00926263
Title: A Phase 1, Open Label Study To Evaluate The Pharmacokinetics, Pharmacodynamics, And Effect On QT/QTc Interval For CP-751,871 Following Single Intravenous Administration To Healthy Adult Subjects
Brief Title: A Pharmacokinetic And QT Study Of CP-751,871 In Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A4021037
Record Dates: First submitted 2009-06-21; First posted 2009-06-23 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Pharmacodynamics; QTc interval prolongation
MeSH Terms: interventions — figitumumab; Moxifloxacin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 mg/kg cohort (Experimental)
  Interventions: Biological: CP-751,871
- 20 mg/kg cohort (Experimental)
  Interventions: Biological: CP-751,871
- 20/20 mg/kg cohort (Experimental)
  Interventions: Biological: CP-751,871, moxifloxacin, saline

INTERVENTIONS:
Biological: CP-751,871 — single dose, 1-hr IV infusion
  Arms: 10 mg/kg cohort
Biological: CP-751,871 — single dose, 1-hr IV infusion
  Arms: 20 mg/kg cohort
Biological: CP-751,871, moxifloxacin, saline — Two doses at 20 mg/kg each on two consecutive days, each administered via 1-hr IV infusion
  Arms: 20/20 mg/kg cohort

SUMMARY:
This study is primarily to evaluate the single dose pharmacokinetics of CP-751,871 and its effect on QT interval prolongation.

DETAILED DESCRIPTION:
This study was terminated on October 30th, 2009. While the study was terminated due to adverse events and altered benefit/risk ratio in healthy subjects, the findings in healthy volunteers are not considered to alter the benefit/risk evaluation of figitumumab in cancer patients. No changes due to the termination of this study are anticipated in the conduct of the ongoing cancer patient studies with figitumumab at this time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or healthy female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* 12-lead ECG demonstrating QTc >450 msec at screening or other clinically significant abnormalities at screening.
* History or family history of risk factors for QTc interval prolongation or torsades de pointes (eg, organic heart disease, congestive heart failure, hypokalemia, hypomagnesemia, congenital long QT syndrome, myocardial ischemia or infarction); family history of sudden death.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021037&StudyName=A%20Pharmacokinetic%20And%20QT%20Study%20Of%20CP-751%2C871%20In%20Healthy%20Subjects%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study participants were planned to be assigned to 1 of 3 sequential dosing cohorts: CP-751,871 at 10 mg/kg; at 20 mg/kg; 2 doses of 20 mg/kg on consecutive days. Dosing was via intravenous (IV) administration. The third dosing cohort (2 doses of 20 mg/kg on consecutive days) did not enroll participants due to early termination of the study.
Groups:
- CP-751,871 10 mg/kg: A single dose of CP-751,871 at 10 mg/kg following an 8 hour fast, administered via 1-hour IV infusion.
- CP-751,871 20 mg/kg: A single dose of CP-751,871 at 20 mg/kg following an 8 hour fast, administered via 1-hour IV infusion.
Period: Overall Study
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Started | 16 | 12
Completed | 16 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg | Total
Number analyzed (Participants) | 16 | 12 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 30.9 (6.3) | 30.3 (7.7) | 30.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 12 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 3 | 7
  Black | 10 | 8 | 18
  Asian | 0 | 1 | 1
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1 pre-dose and 1 hour post-dose, Day 2 (24 hours post-dose), 8, 15, 22, 29, 43, 57, 71 and 85
Population: All treated participants.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
mg/L | 225.1 (54.175) | 420.6 (62.175)

2. Primary Outcome: Area Under the Curve From Time Zero to the Last Time Point With Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Day 1 pre-dose and 1 hour post-dose, Day 2 (24 hours post-dose), 8, 15, 22, 29, 43, 57, 71 and 85
Population: All treated participants.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
mg*h/L | 80740 (14184) | 184000 (27811)

3. Primary Outcome: Plasma Clearance (CL)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Day 1 pre-dose and 1 hour post-dose, Day 2 (24 hours post-dose), 8, 15, 22, 29, 43, 57, 71 and 85
Population: All treated and evaluable participants (had measurements related to the PK parameter stated above).
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 13 | 12
mL/day/kg | 2.808 (0.3804) | 2.353 (0.4346)

4. Primary Outcome: Apparent Volume of Distribution (Vz)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: Day 1 pre-dose and 1 hour post-dose, Day 2 (24 hours post-dose), 8, 15, 22, 29, 43, 57, 71 and 85
Population: All treated and evaluable participants (had measurements related to the PK parameter stated above).
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 13 | 12
mL/kg | 84.89 (13.731) | 92.17 (14.978)

5. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 1 pre-dose and 1 hour post-dose, Day 2 (24 hours post-dose), 8, 15, 22, 29, 43, 57, 71 and 85
Population: All treated and evaluable participants (had measurements related to the PK parameter stated above).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 13 | 12
days | 21.08 (2.9950) | 27.75 (5.7969)

6. Primary Outcome: QTc Using Fridericia's Correction Method (QTcF) After Receiving CP-751,871 at the 20/20 mg/kg Dose Level
Description: QTcF is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole, corrected for heart rate using Fridericia's correction
Time Frame: Day 1 at 1 and 24 hours post-dose, Day 7, 28
Population: Data not obtained due to early termination of the study.
Groups:
- CP-751,871 20/20 mg/kg: Participants not enrolled due to early termination of the study.
Arm/Group | CP-751,871 20/20 mg/kg
Number analyzed (Participants) | 0

7. Secondary Outcome: QTcF After Receiving Moxifloxacin at the Historical Moxifloxacin Median Tmax of 3 Hours
Time Frame: baseline, 3 hours postdose
Population: Data not obtained due to early termination of the study.
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Serum Concentration of Insulin-like Growth Factor 1 (IGF-1)
Description: IGF-1 is one of the IGF-axis related biomarkers. Part of the secondary objectives of the study was to explore the relationships of plasma CP-751,871 concentrations to such biomarkers. Cmax is the mean ± standard deviation (SD) concentration observed at the time of maximal change from baseline.
Time Frame: Day 1 pre-dose (Baseline), 1 hour post dose, Day 2 (24 hours post-dose), Day 8, 15, 22, 29, 43, 57, 71, 85
Population: All treated participants who had at least 1 postdose concentration measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
ng/mL
  Baseline | 138 (33) | 128 (23)
  at Cmax | 566 (142) | 610 (143)

9. Secondary Outcome: Serum Concentration of Free Insulin-like Growth Factor 1 (IGF-1)
Description: as for outcome 8
Time Frame: Day 1 pre-dose, 1 hour post dose, Day 2 (24 hours post-dose), Day 8, 15, 22, 29, 43, 57, 71, 85
Population: All treated participants who had at least 1 postdose concentration measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
ng/mL
  Baseline | 17.2 (6.6) | 13.9 (5.6)
  at Cmax | 143 (45) | 168 (43)

10. Secondary Outcome: Serum Concentration of Insulin-like Growth Factor 2 (IGF-2)
Description: IGF-2 is one of the IGF-axis related biomarkers. Part of the secondary objectives of the study was to explore the relationships of plasma CP-751,871 concentrations to such biomarkers. Cmax is the mean ± standard deviation (SD) concentration observed at the time of maximal change from baseline.
Time Frame: Day 1 pre-dose, 1 hour post dose, Day 2 (24 hours post-dose), Day 8, 15, 22, 29, 43, 57, 71, 85
Population: All treated participants who had at least 1 postdose concentration measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
ng/mL
  Baseline | 1550 (440) | 1476 (229)
  at Cmax | 2039 (582) | 1909 (275)

11. Secondary Outcome: Serum Concentration of Insulin-like Growth Factor Binding Protein 3 (IGFBP-3)
Description: IGFBP-3 is one of the IGF-axis related biomarkers. Part of the secondary objectives of the study was to explore the relationships of plasma CP-751,871 concentrations to such biomarkers. Cmax is the mean ± standard deviation (SD) concentration observed at the time of maximal change from baseline.
Time Frame: Day 1 pre-dose, 1 hour post dose, Day 2 (24 hours post-dose), Day 8, 15, 22, 29, 43, 57, 71, 85
Population: All treated participants who had at least 1 postdose concentration measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
ng/mL
  Baseline | 2041 (546) | 1978 (496)
  at Cmax | 4945 (1035) | 5819 (1310)

12. Secondary Outcome: Serum Concentration of Insulin
Description: Insulin is one of the IGF-axis related biomarkers. Part of the secondary objectives of the study was to explore the relationships of plasma CP-751,871 concentrations to such biomarkers. Cmax is the mean ± standard deviation (SD) concentration observed at the time of maximal change from baseline.
Time Frame: Day 1 pre-dose, 1 hour post dose, Day 2 (24 hours post-dose), Day 8, 15, 22, 29, 43, 57, 71, 85
Population: All treated participants who had at least 1 postdose concentration measurement.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
mIU/mL
  Baseline | 5.13 (3.17) | 4.07 (3.30)
  at Cmax | 37.6 (23.8) | 40.0 (34.5)

13. Secondary Outcome: Serum Concentration of Fasting Glucose
Description: Glucose is one of the IGF-axis related biomarkers. Part of the secondary objectives of the study was to explore the relationships of plasma CP-751,871 concentrations to such biomarkers. Cmax is the mean ± standard deviation (SD) concentration observed at the time of maximal change from baseline.
Time Frame: Day 1 pre-dose, 1 hour post dose, Day 2 (24 hours post-dose), Day 8, 15, 22, 29, 43, 57, 71, 85
Population: All treated participants who had at least 1 postdose concentration measurement.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
mg/dL
  Baseline | 87.7 (6.4) | 87.3 (5.1)
  at Cmax | 104 (21) | 101 (16)

14. Secondary Outcome: Anti-drug Antibodies (ADA) Against CP-751,871 in Serum Samples
Description: Number of participants who tested positive for ADA
Time Frame: Day 1 pre-dose, Day 15, 29, 57, 85
Population: All treated participants.
Measure: Number; unit: number of participants
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 16 | 12
number of participants
  Nominal Day 1 | 0 | 0
  Nominal Day 15 | 0 | 0
  Nominal Day 29 | 0 | 0
  Nominal Day 57 | 0 | 0
  Nominal Day 85 | 0 | 0

ADVERSE EVENTS:
Arm/Group | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 9/16 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 10 mg/kg (N=16) | CP-751,871 20 mg/kg (N=12)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 9
Keratoconjunctivitis sicca (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 9
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 3
Pyrexia (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Chlamydial infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Audiogram abnormal (Investigations) | 2 | 0
Echocardiogram abnormal (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Schirmer's test abnormal (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 3
Paraesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated prior to enrollment of participants into Cohort 3 (2 doses of 20 mg/kg on consecutive days). Therefore, endpoints relating to that cohort were not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.